CLINICAL TRIAL: NCT06885944
Title: Probiotics for Preterm Infants After Full Enteral Feeding
Brief Title: Probiotics for Preterm Infants
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Fuat Emre Canpolat, Professor, Ankara City Hospital Bilkent
Other Study IDs: ABSH-Neo-Pro1
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Preterm Infant Feeding Outcomes; Probiotic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Preterm infants receiving probiotics
  Interventions: Dietary Supplement: Probiotic mix preparation; Dietary Supplement: Bifidobacteria

INTERVENTIONS:
Dietary Supplement: Probiotic mix preparation — Bifidobacterium containing supplement with vitamin D will start after preterm infants reaches full enteral feeding
Dietary Supplement: Bifidobacteria — Rather than early period we will start probiotics after infant receive full enteral feedings

SUMMARY:
Probiotics will be used for preterm infants under 32 weeks of gestation and under 1500 g birthweight. Our aim was to investigate the effects of probiotics for stable preterm infants after extubation and who reached full enteral feeding. There are some hesitations among care-givers to start probiotics early due to safety issues although there are many positive effects of these products reported int the literature.

DETAILED DESCRIPTION:
Our study included premature babies with a birth weight of less than 1500 grams, born at less than 32 weeks of gestation, and without congenital anomalies.

Approval was obtained from the hospital's clinical research ethics committee before starting the study. The decision to start probiotics was made when these premature babies were fully enteral fed. The study design was created as a cohort and case-control study (No randomisation). When clinicians decided to start probiotic support for premature babies with good general health and no additional problems, probiotics were added to the baby's order.

ELIGIBILITY:
Inclusion Criteria: <32 weeks, <1500 g birthweight -

Exclusion Criteria: Congential anomalies, still parenteral feeding, BW<800 gr and <23 weeks of GA

-

Ages: 7 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: preterm infants with a gestational age lower than 32 weeks and 1500 g of birthweight, reached to fully enteral feeds
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-30 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Antropometric measures | 2 months
  daily weight gain mg/kg/day

SECONDARY OUTCOMES:
Metabolic profile | 2 months
  Ca, P, ALP, Urea and biochmeical markers for nutritional status

CONTACTS AND LOCATIONS:
Overall Officials: FUAT EMRE CANPOLAT, MD, Principal Investigator — Ankara City Hospital Bilkent

IPD SHARING:
Plan to Share IPD: Undecided